CLINICAL TRIAL: NCT04515914
Title: Clinical Relevance of DNA Methyltransferase and Histone Deacetylase Gene Single Nucleotide Polymorphism in Myelodysplastic Syndrome
Brief Title: Clinical Relevance of DNMT and HDAC Gene SNP on the Response to Decitabine Therapy for Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan (Dennis) Kim/Assistant professor, Samsung Medical Center
Other Study IDs: 2009-04-012
Record Dates: First submitted 2010-06-02; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2011-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: DNA methyltransferase gene; Histone deacetylase gene; Single nucleotide polymorphism; Decitabine; Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples from MDS patients receiving Decitabine therapy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Decitabine therapy: The patients are treated with decitabine at least 1 cycles
- non-Decitabine therapy: The Patients are diagnosed as MDS and do not be treated with decitabine therapy

SUMMARY:
Recent investigations have demonstrated that DNMT gene polymorphisms can contribute to the inter-individual variants in DNMT expression. Accordingly, we hypothesized that the DNMT and HDAC genes SNPs could predict the outcomes of decitabine therapy for myelodysplastic syndrome. Prospective collection of DNA from peripheral blood will be performed in the patients with MDS before commencement of decitabine therapy. We will evaluate the efficacy decitabine therapy according to the DNMT or HDAC gene SNPs in terms of following parameters: 1) hematolotic response (HR) or improvement (HI), or requirement of decitabine dose to achieve HR or HI, 2) complete (CR) or partial response (PR), or requirement of decitabine dose to achieve CR or PR, and 3) time to relapse or progression of MDS.

The objective of this study is 1) to determine genotypes from DNA samples from MDS patients receiving Decitabine therapy, 2) to determine the association of clinical outcomes (HR, HI, CR, PR or time to progression to leukemia) following decitabine therapy with DNMT or HDAC genotypes, and 3) to analyze the impact of cytogenetic risk on the response or leukemic evolution following decitabine therapy for MDS.

DETAILED DESCRIPTION:
This study will include the patients who signed the subject informed consent form among the patients with MDS who were chosen to be treated with Decitabine (Part I), plus additional 140 MDS patients as a historical control (Part II). Approximately, 68 patients will be included who satisfy the following inclusion and exclusion criteria in the Part I study.

Prospective collection of DNA from peripheral blood will be performed in the patients with MDS before commencement of decitabine therapy. We will evaluate the efficacy decitabine therapy according to the DNMT or HDAC gene SNPs in terms of following parameters: 1) hematolotic response (HR) or improvement (HI), or requirement of decitabine dose to achieve HR or HI, 2) complete (CR) or partial response (PR), or requirement of decitabine dose to achieve CR or PR, and 3) time to relapse or progression of MDS.

Genotyping will be undertaken using the Sequenom® iPLEX platform™, according to the manufacturer's instructions (www.sequenom.com; Sequenom Inc, San Diego, CA, USA). Whole blood samples will be obtained according to the declaration of Helsinki. DNA will be extracted using the Puregene DNA purification Kit (Gentra Systems Inc, Minneapolis, MN, USA). The detection of SNPs will be performed by the analysis of primer extension products generated from previously amplified genomic DNA using a Sequenom chip-based matrix-assisted laser desorption / ionization time-of-flight (MALDI-TOF) mass spectrometry platform. Multiplex SNP assays will be designed using SpectroDesigner software (Sequenom). Ninety-six well plates containing 2.5 ng DNA in each well will be amplified by PCR following the specifications of Sequenom. Unincorporated nucleotides in the PCR product will be deactivated using shrimp alkaline phosphatase. Allele discrimination reactions will be conducted by adding the extension primer(s), DNA polymerase, and a cocktail mixture of deoxynucleotide triphosphates and di-deoxynucleotide triphosphates to each well. MassExtend clean resin (Sequenom) will be added to the mixture to remove extraneous salts that could interfere with MALDI-TOF analysis. The primer extension products will be then cleaned and spotted onto a SpectroChip. Genotypes will be determined by spotting an aliquot of each sample onto a 384 SpectroChip (Sequenom), which is subsequently read by the MALDI-TOF mass spectrometer.

All statistical tests will be two-sided with the significance level set as 0.05 unless otherwise stated. The statistical data will be obtained using an SAS version 9.1 (SAS Institute, Cary NC, USA). Followings are the endpoints for the study.

1. Primary endpoint evaluation data

   • Response rate: A response rate will be obtained and its confidence interval estimated to be evaluated through chi-square test. If the main endpoints which may influence the final evaluation must be controlled, stratified analysis (Cochran-Mantel-Haenzel, etc.) will be conducted. If all the subjects' characteristic endpoints must be controlled, the logistic regression model will be used for analysis.
2. Secondary endpoint evaluation data

   * Overall survival: survival will be evaluated from the registration day to death through Kaplan-Meier method.
   * Progression free survival: : The time of progression from MDS to AML and death from any cause. Progression free survival will be analyzed through Kaplan-Meier method.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Decitabine treatment group

      * Male and female aged 18 years or older.
      * The patients diagnosed with (primary or secondary) MDS
      * Patients with an IPSS score of ≥ Int-1
      * Patients treated with Decitabine at least 1 cycles.
      * Signed and dated informed consent before the start of genetic study using genomic DNA derived from blood sample.
   2. Historical control group

      * Male and female aged 18 years or older.
      * The patients diagnosed with (primary or secondary) MDS
2. Exclusion Criteria:

   * Patients diagnosed with acute myelogenous leukemia (AML, bone marrow stem cell counts exceeding 20%) or other progressive malignant diseases.
   * Diagnosis of chronic myelomonocytic leukemia (CMML) or MDS/MPD excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include the patients who signed the subject informed consent form among the patients with MDS who were chosen to be treated with decitabine, plus additional MDS patients as a historical control.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 18 months

SECONDARY OUTCOMES:
Time to progression or hematologic improvement | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D.,Ph.D., Principal Investigator — Division of Hematology and Oncology/Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea